CLINICAL TRIAL: NCT03074838
Title: Reduced Inflammatory Response Using Transcatheter Aortic Valve Replacement as Compared to Conventional Surgery
Brief Title: Inflammatory Response to Aortic Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Erik Fosse, Head of Department, Professor, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/7919
Record Dates: First submitted 2017-02-28; First posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Aortic Valve Stenosis
Keywords: Cardiac surgery; TAVI
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: A case Control study were patients undergoing two surgical Methods for aortic valve repair is compared
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transarterial aortic valve implantation (Experimental): Patients that are treated by trans arterial valve implantation (TAVI)
  Interventions: Procedure: Transarterial aortic valve implantation - TAVI
- Surgical aortic valve replacement (Active Comparator): Patients that are treated by surgical aortic valve replacement (SAVR)
  Interventions: Procedure: Surgical aortic valve replacement - SAVR

INTERVENTIONS:
Procedure: Transarterial aortic valve implantation - TAVI — After insertion of a guidewire, either through the femoral artery or through the ascending aorta, the aortic ostium is dilated by a balloon and the valve is introduced through a catheter and expanded in the ostium.
  Arms: Transarterial aortic valve implantation
Procedure: Surgical aortic valve replacement - SAVR — The patient is operated through a sternotomy and coupled to a heart lung machine. The aorta is opened and the native valve excised. Then a biological artificial heart valve is sutured in place.
  Arms: Surgical aortic valve replacement

SUMMARY:
A controlled un-randomized trial where the inflammatory response in 18 patients admitted for TAVI procedure is compared to the inflammatory response in 18 patients admitted for conventional surgical valve replacement. Clinical outcomes are recorded and compared between the Groups. As a secondary endpoint, the inflammatory response was also compared between the patients receiving either transfemoral or trans aortal TAVI.

DETAILED DESCRIPTION:
18 patients admitted successively for conventional surgical aortic valve replacement and 18 patients admitted for transcatheter aortic valve implantation (TAVI) (9 transfemoral and 9 transaortic) are included.

A plasma sample is obtained at defined timepoints before, during and after surgery. At each time points the following biomarkers are analyzed:Concentrations of the complement activation products C3bc and the terminal C5b-9 complement complex (TCC), the neutrophil release product myeloperoxidase (MPO), the cytokines IL-6, eotaxin, MCP-1 and MIP-1β (12). As marker of a myocardial cellular injury troponin T levels will be analyzed. The following clinical outcomes will also be monitored: Death (in hospital, 30 day and one year), blood transfusion, stroke, myocardial infarction.

A dedicated registry will be established at the hospital according to the hospital's standard for storage of patient data. The registry will be deleted after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for aortic valve replacement without need for concurrent surgery

Exclusion Criteria:

* known inflammatory disease and anti-inflammatory treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Generation of several inflammatory markers measured through repeated blood samples | 24 hours
  The total generation of several inflammatory markers is compared between the groups

SECONDARY OUTCOMES:
Blood loss | 24 hrs
  ml blood loss compared between the groups
Blood transfusion | 24 hrs
  Number of blood Products tranfused after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Erik Fosse, MD PhD, Principal Investigator — Oslo University Hospital/University of Oslo; Karoline KH Fiane, Med Student, Study Chair — University of Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fiane KKH, Dahle G, Bendz B, Halvorsen PS, Abdelnoor M, Mollnes TE, Fosse E. Reduced inflammatory response by transcatheter, as compared to surgical aortic valve replacement. Scand Cardiovasc J. 2018 Feb;52(1):43-50. doi: 10.1080/14017431.2017.1416157. Epub 2017 Dec 12. PMID 29233022